CLINICAL TRIAL: NCT02700217
Title: Does Adding Spinal Anaesthesia to a General Anaesthetic Technique Influence Readiness for Discharge in Patients Having Hand Assisted Laparoscopic Live Donor Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R04134
Record Dates: First submitted 2016-02-09; First posted 2016-03-07 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Surgery
Keywords: Donor Nephrectomy
MeSH Terms: interventions — Bupivacaine; Heroin; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Anaesthesia (Experimental): 2.5ml of heavy 0.5% Bupivacaine, 400mg of Diamorphine (Spinal Anaesthesia) & IV infusion of Remifentanil 0.2-0.3ug/kg/min, Propofol 2-3mg/kg and 0.2 mg/kg of Cistracurium (General Anaesthesia)
  Interventions: Procedure: Bupivacaine and Diamorphine; Procedure: Remifentanil, Propofol and Cistracurium
- Rectus Sheath Injection (Active Comparator): 50ml of 0.25% I-Bupivacaine max 2mg/kg (IV block Anaesthesia) injected into rectus sheath bilaterally & IV infusion of Remifentanil 0.2-0.3ug/kg/min, Propofol 2-3mg/kg and 0.2 mg/kg of Cistracurium (General Anaesthesia)
  Interventions: Procedure: Remifentanil, Propofol and Cistracurium; Procedure: Bupivacaine and Rectus Sheath injection

INTERVENTIONS:
Procedure: Bupivacaine and Diamorphine
  Arms: Spinal Anaesthesia
Procedure: Remifentanil, Propofol and Cistracurium
Procedure: Bupivacaine and Rectus Sheath injection
  Arms: Rectus Sheath Injection

SUMMARY:
About 1100 living donor nephrectomies are performed in the UK every year contributing to almost 35% of all the kidney transplants. Laparoscopic surgical techniques are general employed for donor nephrectomy as they are associated with a shorter hospital stay and faster return to normal physical functioning. Local anaesthetic infiltration technique with or without spinal anaesthesia in combination with a general anaesthetic is increasingly being used as part of enhanced recovery programme across general surgery. The impact of combined spinal and general anaesthesia along with local infiltration and rectus sheath blocks on acute pain has not been studied in patients undergoing hand assisted laparoscopic live donor nephrectomy.

The investigators plan to investigate whether adding a spinal anaesthetic to a conventional general anaesthetic technique actually influences clinical outcomes of length of hospital stay and acute pain in patients undergoing hand assisted laparoscopic live donor nephrectomy.

The investigators plan to randomise 90 patients undergoing hand assisted laparoscopic live donor nephrectomy over 24 month period at Central Manchester University hospitals and divide them in two groups of 45 each. Group A will receive a general anaesthetic (GA) with spinal anaesthesia (Spinal group) and Group B will receive a GA with a rectus sheath block (Rectus sheath group) and local anaesthetic infiltration

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 status
* Patients aged between 18-65 years

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Allergy to bupivacaine
* Patients who have had previous abdominal surgery
* Patients having chronic pain or any medications for chronic pain
* Any patient in whom spinal anaesthesia is contra-indicated
* Patients on anti-platelet or anti-thrombotic therapy.
* Patient requiring interpreter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Assessment of readiness for discharge from hospital to determine Length of stay, after renal surgery, using a blinded Nurse assessment of patient. | 5 days
  From Day 2 a nurse blinded to both groups will assess the readiness for discharge at 10:00, 14:00 and at 18:00 hours. The patient would be considered suitable for discharge if the following criteria are met:
  (i) Able to get in and out of bed, (ii) Able to get dressed, (iii) Able to go to toilet without walking aids, (iv) Pain manageable with oral analgesics, (v) Patient willing to be discharged.
  Length of stay (LOS) would be calculated as the time from the end of surgery until the subject met the discharge criteria from the ward. The actual day and time the patient leaves the hospital would be noted as well.

SECONDARY OUTCOMES:
Assessment of Pain from surgery to discharge tested at intervals using an 11 point linear numerical rating scale utilised for assessment of pain. | 5 days
  Pain scores at rest and on movement along with PONV scores with anti-emetics will be assessed thrice daily at 10:00, 14:00 and 18:00 on Day 1. Total oxycodone consumption in the first 24 hours after surgery will be noted.
  In the ward, the pain scores at rest and at movement would be assessed at 3, 6, 12 and 24 hours from the end of surgery using the NRS scoring system by a nurse who would be blinded to both the groups.
The total patient controlled analgesia (PCA) morphine consumption | 5 days
Assessing the side effects of the anaesthetic technique specifically looking at PDPH throughout the recovery process in hospital, using the PONV | 5 days
  Assessing the side effects of the anaesthetic technique specifically looking at vasopressor use peri-operatively, postoperative nausea and vomiting, post dural puncture headache (PDPH) and urinary re-catherisation rates throughout the recovery process in hospital, using the Postoperative nausea and vomiting scale (PONV).
Assessing the side effects of the anaesthetic technique specifically looking at PDPH throughout the recovery process in hospital, using the VAS | 5 days
  Assessing the side effects of the anaesthetic technique specifically looking at vasopressor use peri-operatively, postoperative nausea and vomiting, post dural puncture headache (PDPH) and urinary re-catherisation rates throughout the recovery process in hospital, using the Visual analogue Scale (VAS) for nausea anchored with 'no nausea' and 'worst possible nausea'.
Assessment of Patient Satisfaction using the Patient Anaesthesia Satisfaction Scale (PASS) | 5 days
  Before leaving the hospital, all patients would be asked to rate the anaesthesia and the pain relief they had received on a 100 mm scale where 0=worst imaginable experience and 100 =best possible experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Bhatia K, Columb M, Wadsworth R, Macnab W, Jepegnanam C, Campbell T, Van Dellen D. Effect of rectus sheath block vs. spinal anaesthesia on time-to-readiness for hospital discharge after trans-peritoneal hand-assisted laparoscopic live donor nephrectomy: A randomised trial. Eur J Anaesthesiol. 2021 Apr 1;38(4):374-382. doi: 10.1097/EJA.0000000000001337. PMID 33009185